CLINICAL TRIAL: NCT00629525
Title: A Single Arm, Two Center, Phase II Study of RAD001 in Patients With Metastatic, Hormone-Refractory Prostate Cancer
Brief Title: RAD001 in Patients With Metastatic, Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel George, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009495; 7521 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Hormone Refractory Prostate Cancer
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): RAD001 at a dose of 10 mg PO daily
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 at a dose of 10 mg PO daily
  Other Names: Everolimus

SUMMARY:
The purpose of this study is to determine the biochemical response rate (PSA) to single agent RAD001 in patients with metastatic hormone-refractory prostate cancer (HRPC).

DETAILED DESCRIPTION:
This is a single center, Phase II study of RAD001 in men with HRPC. The study design is a straight forward, two-stage design with tumor biopsies scheduled at screening and again at 4 weeks. FLT-PET scans are performed at screening and again at day 28, following initiation of treatment in the first 10 patients. Patients are assessed for adverse events every two weeks for the first month and monthly thereafter. Patients are assessed for response by PSA every 4 weeks and when applicable, for objective response every 2 months. If 4 or more responses are seen in the first 39 patients then the study will expand to 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate
* Clinical or radiographic evidence of metastatic disease
* ADT using LHRH agonist (eg leuprolide, goserelin) must continue on therapy. However, ketoconazole, estrogens, and all other forms of hormonal manipulation are not permitted on study.
* Evidence of disease progression on ADT as evidenced by:

  * 2 consecutive PSA levels 50% or greater above the PSA nadir achieved on ADT and separated at least 1 week apart, or
  * Radiographic evidence of disease progression defined by RECIST criteria and compared to prior studies on ADT.
* A minimum of 6 weeks has elapsed off of anti-androgen therapy without withdrawal response.
* A minimum of 4 weeks from any prior radiation therapy, surgery, chemotherapy or other investigational agent
* Biopsies will not be performed if platelet counts < 75,000/ ul, PTT, PT or INR > 1.4 times control
* Patients must have normal organ and marrow function as defined below:
* hemoglobin > 9.0g/dL
* absolute neutrophil count > 1,500/μl
* platelets > 100,000/μl
* total bilirubin < 1.5 X upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) < 2.5 X ULN
* creatinine < 1.5 X ULN
* total fasting cholesterol < 350
* total triglycerides < 300
* Patients on antilipid therapy may participate in this study.
* Age > 18 years
* ECOG performance status 0 or 1
* Ability to swallow and retain oral medication
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of solid organ or stem cell transplantation
* Also, no current use of chronic immunosuppressive therapy is allowed
* Patients with known brain metastases (or history of brain metastases)
* History of HIV, hepatitis B, or hepatitis C infection
* Patients who have received investigational, biologic, hormonal (other than ADT), immunotherapy, or chemotherapy less than 4 weeks prior to entry on this study or have not recovered from the toxic effects of such therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (requiring antifungal, antibiotic or antiviral therapy), symptomatic congestive heart failure (NYHC III or greater), unstable angina pectoris, cardiac arrhythmia (uncontrolled SVT or any VT), or psychiatric illness/social situations that would limit compliance with study requirements
* History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism or excretion of study drugs.
* Any unresolved bowel obstruction or diarrhea

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-08; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J George, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University MEdical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001
Started | 35
Completed | 32
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 71 [52 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response Rate
Description: Number of participants with 50% decline in serum PSA from baseline was pre-set as the primary measure of disease response.
Time Frame: Patients were followed for a median of 315 days
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 35
participants | 0

2. Secondary Outcome: Pathologic Response
Description: Number of participants with either a 50% or greater decrease in proliferation index or a 50% or greater increase in apoptotic index
Time Frame: Patients were followed for a median of 315 days
Population: Only subjects with paired samples were included in this analysis
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 4
participants | 0

3. Secondary Outcome: Progression Free Survival
Description: Time in months from the start of study treatment to the date of first progression according to RECIST 1.0, or to death due to any cause. Patients alive who had not progressed as of the last follow-up had PFS censored at the last follow-up date. Median PFS was estimated using a Kaplan-Meier curve.
Time Frame: Patients were followed for a median of 315 days, with the last patient censored at 1309 days.
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001
Number analyzed (Participants) | 35
months | 3.58 [2.07 to 4.83]

4. Secondary Outcome: Molecular Response
Description: Functional extent of mTOR inhibition by changes in the phosphorylation status of pS6 in prostate tumors.
Time Frame: Patients were followed for a median of 315 days
Population: Immunohistochemistry (IHC) for pS6 was compared for 9 pairs of samples for which paraffin embedded tissue was available.
Measure: Mean (Full Range); unit: percentage of decrease
Arm/Group | RAD001
Number analyzed (Participants) | 9
percentage of decrease | 60.11 [14.29 to 100.00]

5. Secondary Outcome: Clinical Response
Description: The percentage of participants with a complete or partial response as defined by RECIST 1.0. Response Criteria are defined below:
  Complete Response: Disappearance of all target lesions Partial Response: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD
Time Frame: Patients were followed for a median of 315 days
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 35
participants | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: data were collected in Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and converted to version 4.0 for Clinicaltrials.gov entry
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 8/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=35)
Myocardial infarction (Cardiac disorders) | 1
Death NOS (General disorders) | 2
Sepsis (Infections and infestations) | 1
INR increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Nervous system disorders - spinal cord compression (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=35)
Anemia (Blood and lymphatic system disorders) | 14
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 11
Dry Mouth (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify: Mucositis (Gastrointestinal disorders) | 19
Mocositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 10
Chills (General disorders) | 2
Edema Limbs (General disorders) | 2
Fatigue (General disorders) | 18
Facial Pain (General disorders) | 5
Fever (General disorders) | 5
Non-cardiac chest pain (General disorders) | 2
Alanine aminotransferase increased (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 15
Cholesterol high (Investigations) | 11
Creatinine increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 17
Weight loss (Investigations) | 11
White blood cell decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 17
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 17
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes